CLINICAL TRIAL: NCT07094217
Title: Fluoroless Conduction System Implant
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 23HH8384
Record Dates: First submitted 2025-07-17; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pacemaker; Conduction System Pacing
Keywords: fluoroless; conduction system pacing; left bundle area pacing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Derivation: These patients will undergo the research protocol. In these patients, we will attempt to implant a permanent conduction system pacing lead, in lieu of the RV or LV lead. The lead will be implanted by operators who have implanted more than 40 leads to overcome the learning curve.
- Validation: An optimised work flow will be derived using the information collected from the derivation cohort. Namely, the target areas for FAM and electro-anatomical maps will be determined, and the successful pattern of lead septum interaction on CARTO will be defined.
  The streamlined workflow will then be applied to 25 prospective patients. The success rates, procedure time, fluoroscopy time, capture threshold, number of attempted lead deployments and complication rates will be assessed.
- Control: The control arm will consist of 25 patients undergoing a conduction system pacemaker using conventional pacing methods, with the same pacing indications as the study arm

SUMMARY:
Conduction system pacing is a new way of stimulating the heart using pacemaker wires. Traditional pacemakers stimulate the heart muscle which causes disordered heart beats: the walls of the heart move at different times. This wears down the heart over time.

Conduction system pacemakers stimulate the heart's electrical system directly producing natural heart beats that are much less disordered. These pacemakers can be challenging to insert with different heart shapes, sizes and scars. This can increase procedure times and time exposed to xray as pacemakers are inserted using x-rays to guide where the lead is implanted.

This study aims to allow conduction system pacemakers to be implanted without the use of normal xray (fluoroscopy).

The investigators will create an anatomical shell of the heart using special plastic (mapping) catheters that is inserted within the heart from the groin. The investigators will use a special heart scanning (echo) catheter to see how the pacemaker wire is inserted into the heart muscle. The investigators will use MRI to confirm that the information we collect is accurate. Using this information the investigators will create a protocol to implant a lead that does not require xray, using only the mapping catheter.

DETAILED DESCRIPTION:
A total of 75 patients will be recruited for the study

50 patients with a ventricular pacing indication (high grade atrioventricular block and symptomatic trifasicular or bifasicular block) for pacing will be recruited prospectively. The patients will be divided into two groups; 25 patients in the derivation cohort and 25 patients in the validation cohort. The derivation cohort will undergo a detailed research protocol to determine the optimised work flow and this will be applied prospectively to the validation cohort.

The success rates, procedure times, complication rates and fluoroscopy times will be assessed. The 25 patients undergoing conventional methods of conduction system pacing will be recruited as a control arm to compare these outcomes.

In summary, the 75 patients will be grouped as following; 25 patients in the derivation cohort, 25 patients in the validation cohort and 25 patients in the control arm.

Methodology

Derivation The derivation cohort will comprise of 25 prospectively recruited patients. These patients will undergo the research protocol. In these patients, the investigators will attempt to implant a permanent conduction system pacing lead, in lieu of the RV or LV lead. The lead will be implanted by operators who have implanted more than 40 leads to overcome the learning curve.

Pre-implant Prior to the procedure, patients will undergo a clinically indicated Cardiac MRI. The investigators will use these scans to retrospectively assess for the presence of potential mechanisms which could prevent successful lead implantation, such as the presence of septal fibrosis and chamber dimensions, so that we can assess how these can contribute to challenges at the time of implant. We will also be able to review mechanisms for successful implants. This information will be corroborated with data collected from the electro-anatomical maps.

The MRI scans will also be used to merge the anatomical information using CartoMerge to reduce procedure times by building the anatomical geometry prior to the mapping-catheter collecting this information invasively.

During Implant

The participants will undergo the following procedural steps after written informed consent is gained:

1. A left infraclavicular incision and axillary access for the lead will be gain as per standard clinical protocol.
2. Access from the femoral vein will be sought where a sheath will be placed in the femoral vein to introduce the mapping catheter.
3. Fast anatomical mapping (FAM) of the right atrial and right ventricular anatomy will be made where CartoMerge has not already created this anatomy. This will include the right ventricle, the tricuspid valve and the right ventricular outflow tract. Activation and voltage maps will be then be made of the His-bundle area (including the His cloud), right ventricle, right ventricular outflow tract and right ventricular septum.

This will help determine a few key aspects

1. Level of conduction system block and therefore guide site of lead deployment
2. Anatomy of the right heart and overcome challenges this may propose
3. Evidence of septal fibrosis and/or scar that need to be overcome
4. Activation pattern of the septum in conduction system block

4. Anatomical FAM maps, voltage maps and activation patterns will be compared against the data collected from the cardiac MRI to assess;

1. Accuracy of anatomy
2. Fibrosis and scar patterns

The CartoMerge module will be used to expedite anatomical mapping using the MRI data collected.

5. The mapping catheter will be removed and an intracardiac echo (ICE) catheter, will be inserted through the femoral vein.

6. The conduction system pacing lead will be inserted through the axillary vein. A right atrial lead will be inserted into the right ventricular apex for back up pacing in the instance the conduction system is bumped. The basal-septum, mid-septum, high-septum and anterior walls will be paced to identify electrical markers for optimal implant sites.

7. The lead will be visualised on the CARTO maps created.

8. The lead will be deployed at the predetermined target site under direct visualisation using the ICE catheter. Through direct visualisation, three key determinants can be assessed:

1. Lead trajectory through the septum with the goal of achieving perpendicularity
2. Lead septum interaction and whether there is evidence of entanglement preventing lead progression.
3. Relationship between the sheath and lead that can lead to or prevent failure of lead deployment.

9. Once the conduction system lead is secured the right atrial lead will be pulled back and secured in the right atrium.

10. The procedure will be completed as per standard clinical implant protocol with routine clinical follow-up thereafter:

The information from echocardiography will be corroborated with the lead-septum interaction visualised on electro-anatomical maps created on CARTO.

In this cohort of patients, the conduction system lead will initially pace the His-bundle then the left bundle in order to collect data for both methods of physiological pacing. The information collected from ICE and electro-anatomical mapping will be used to develop a streamlined workflow that will map targeted areas, where challenging implant sites will be rapidly identified (such as areas of scar), reducing the number of attempted lead deployments and visualise lead-septum interaction, apposition and progression, improving safety parameters.

At the end of the procedure, the lead position will be documented with a very short, single fluoroscopic acquisition. This remains integral for future comparison in the instances of lead complications and in particular lead displacement.

Validation

25 patients will be recruited to the validation cohort.

An optimised work flow will be derived using the information collected from the derivation cohort. Namely, the target areas for FAM and electro-anatomical maps will be determined, and the successful pattern of lead septum interaction on CARTO will be defined.

The streamlined workflow will then be applied to 25 prospective patients. The success rates, procedure time, fluoroscopy time, capture threshold, number of attempted lead deployments and complication rates will be assessed.

Control Arm The control arm will consist of 25 patients undergoing a conduction system pacemaker using conventional pacing methods, with the same pacing indications as the study arm.

Follow-up All 75 patients will have standard clinical follow-up at 6 weeks, 6 months and 1 year. The clinical information at these visits will be used to identify complications rates that will include lead displacement, rise in capture threshold and lead injury, device related infections.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a ventricular pacing indication: high grade atrioventricular block and symptomatic trifasicular, bifasicular block or left bundle branch block LBBB for cardiac resynchronisation therapy
2. Adults willing to take part (ages 18 - 100 years old)
3. Able to give consent.

Exclusion Criteria:

1. Unable to give consent
2. Children age < 18 years and adults > 100 years old
3. Pregnant patients • As per standard of care, female patients of child-bearing age will have a urine pregnancy test prior to their procedure.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients referred for a cardiac pacemaker at Imperial College Healthcare Trust.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Successful conduction system lead implantation with a fluoroless implant protocol | From time of first patient recruited to the last patient recruited in the in the derivation cohort, upto 52 weeks
  The primary objective of this study is to develop a fluoroless implant protocol of conduction system leads using 3D electroanatomical mapping. Electroanatomical mapping will be used to understand the cardiac anatomy, removing the reliance on fluoroscopy to position the pacemaker lead. Successful conduction system lead implant rates will be assessed against a control arm utilising conventional fluoroscopic methods.

SECONDARY OUTCOMES:
Change in fluoroscopy time | From time of first patient recruited to the time of last patient recruited in the validation cohort upto 52 weeks
  Is there a change in the overall procedure and fluoroscopy time with utilisation of targeted lead deployment.
Change in complication rates | From time of first patient recruitment to the 1 year after last patient recruited
  With better visualisation of the cardiac anatomy using the electroanatomical mapping, is there a change in complication rates

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Whinnett, BM.BS, Principal Investigator — Imperial College London, Imperial College Healthcare Trust

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT07094217/Prot_000.pdf